CLINICAL TRIAL: NCT00352261
Title: An Open-Label, 2-Way Crossover Study of Steady-State Intragastric pH Control Comparing 2 Dosage Regimens of Esomeprazole and Lansoprazole in Barrett's Esophagus Patients
Brief Title: An Open Label pH Comparison of Esomeprazole and Lansoprazole in Barrett's Esophagus Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00082
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Esomeprazole; Lansoprazole

INTERVENTIONS:
Drug: Esomeprazole
Drug: Lansoprazole

SUMMARY:
The purpose of the study is to compare the treatment of esomeprazole 40 mg once daily and lansoprazole 30 mg once daily in controlling intragastric pH in Barrett's Esophagus patients

ELIGIBILITY:
Inclusion Criteria:

* Documented history (within 2 yrs of histologically proven BE;
* Aged 18-70 (inclusive);
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Signs of clinically significant GI bleeding within 3 days prior to randomization;
* History of gastric or esophageal surgery;
* Clinically significant illness within 2 weeks prior to first dose of study drug or during study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2006-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Compare pharmacodynamic efficacy of esomeprazole 40 mg & lansoprazole 30 mg once daily in controlling intragastric pH in Barrett's Esophagus patients by evaluation of the percentage of time that intragastric pH is >4.0 over a 24 hr period steady state

SECONDARY OUTCOMES:
Compare pharmacodynamic efficacy of esomeprazole 40 mg & lansoprazole 30 mg bid in controlling intragastric pH in BE patients by evaluation of the % of time intragastric pH is >4.0 over 24 hr period at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Debra Silberg, MD, Study Director — AstraZeneca
Locations (12):
- United States (12):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, North Chicago, Illinois
  - Research Site, Rochester, Minnesota
  - Research Site, Kansas City, Missouri
  - Research SIte, Springfield, Missouri
  - Research Site, Butte, Montana
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Norfolk, Virginia